CLINICAL TRIAL: NCT05651503
Title: The Effect of Oral Probiotics on Oral Hygiene and Halitosis in Orthodontic Patients: a Randomized Controlled Trial
Brief Title: The Effect of Oral Probiotics on Oral Hygiene and Halitosis in Orthodontic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: Align Technology, Inc. (Industry)
Responsible Party: Principal Investigator, Iosif Sifakakis, assistant professor, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444/27.07.2020
Record Dates: First submitted 2022-12-02; First posted 2022-12-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Halitosis; Probiotics; Orthodontic Appliance Complication
Keywords: Halitosis; Probiotics; Fixed Appliances; Aligners
MeSH Terms: conditions — Halitosis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This trial is designed as a prospective, randomized, placebo-controlled, double (investigator and patient) blinded, with four parallel groups and an equal allocation ratio in all groups. In this dose study, the intervention consists of delivery of oral probiotics Lactobacillus Salivarius or placebo lozenges.
  Equal number of males and females will be allocated to each group. In our study oral probiotics Lactobacillus salivarius Oral S1 11 (Prodilac Oral, Frezyderm) will be tested in two different groups:
  Experimental group 1: patients, age 12-18, conventional brackets, Oral probiotics lozenges Experimental group 2: patients, age ≥18, Invisalign™ appliances, Oral probiotics lozenges Control group 1: patients, age 12-18, conventional brackets, placebo lozenges Control group 2: patients, age ≥18, Invisalign™ appliances, placebo lozenges
Who Masked: Participant, Investigator
Masking Description: Two random sequences will be obtained for each age group from www.random.org (2 for patients 12-18 yo and 2 for patients ≥18 yo), one for males and one for females in each age group. Each sequence will be a random ordering of a list of 30 'Ex's and 30 'Co's (Ex: Probiotic, Co: Placebo). The sequence values will be written on standard-sized pieces of paper using a pencil and sealed in opaque numbered envelopes (sequentially numbered from F1 to F30 (female group) and M1 to M30 (male group)) for each group by a person not involved in the project.
  The different lozenges will be labeled 1 or 2 by the manufacturer. The packaging, appearance and taste of lozenges in both intervention and control groups will be identical.
  Clinical measurements of plaque accumulation, gingival inflammation and VSCs levels will be conducted by an assessor blind to treatment allocation. Due to the nature of the intervention, participants and patients can be blinded to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1: patients, age 12-18, conventional brackets, Oral probiotics lozenges (Experimental): 30 patients, age 12-18,with conventional brackets,will get Oral probiotics lozenges
  Interventions: Dietary Supplement: Probiotics
- Experimental group 2: patients, age ≥18, Invisalign™ appliances, Oral probiotics lozenges (Experimental): 30 patients, age ≥18, Invisalign™ appliances,wil get Oral probiotics lozenges
  Interventions: Dietary Supplement: Probiotics
- Control group 1: patients, age 12-18, conventional brackets, placebo lozenges (Placebo Comparator): 30 patients, age 12-18, conventional brackets,will get placebo lozenges
  Interventions: Dietary Supplement: Placebo tablet
- Control group 2: patients, age ≥18, Invisalign™ appliances, placebo lozenges (Placebo Comparator): 30 patients, age ≥18, Invisalign™ appliances,will get placebo lozenges
  Interventions: Dietary Supplement: Placebo tablet

INTERVENTIONS:
Dietary Supplement: Probiotics — In our study oral probiotics Lactobacillus salivarius Oral S1 11 (Prodilac Oral, Frezyderm) will be tested in two Experimental groups
  Arms: Experimental group 1: patients, age 12-18, conventional brackets, Oral probiotics lozenges; Experimental group 2: patients, age ≥18, Invisalign™ appliances, Oral probiotics lozenges
Dietary Supplement: Placebo tablet — In order to avoid possible bias, probiotics will be compared with placebo lozenges/no probiotic in two Control groups
  Arms: Control group 1: patients, age 12-18, conventional brackets, placebo lozenges; Control group 2: patients, age ≥18, Invisalign™ appliances, placebo lozenges

SUMMARY:
Brackets, bands, ligatures and wires in patients receiving orthodontic treatment with fixed appliances are areas that trap food and impede oral hygiene. An ecological environment facilitating the growth of microorganisms (Actinobacillus, Bacteroides, Prevotella etc.) emerges in the mouth and may cause caries, enamel white spots, gingival inflammation and halitosis. Despite the use of specialized orthodontic brushes, interdental brushes, mouthwashes and topical fluorides, plaque removal remains inadequate in patients with fixed orthodontic appliances. On the other hand, patients undergoing orthodontic treatment with aligners have been found to have better oral hygiene because of less plaque accumulation in their mouth.

Probiotics are defined as non-pathogenic bacteria that can benefit the host's general health when taken in sufficient amounts through nutrition. Nowadays probiotics can be used to enhance oral health as they are found to reduce dental bioﬁlm formation, prevent and decrease halitosis in children, adolescents and adults. To date, there are few randomized controlled trials (RCTs) examining the efﬁcacy of oral probiotics in patients with fixed orthodontic appliances and none reporting the incidence of halitosis and the effect of probiotics in orthodontic patients wearing aligners.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of the oral probiotic Lactobacillus salivarius on oral hygiene indices and halitosis in patients wearing orthodontic braces and patients wearing orthodontic aligners. The study is a prospective, randomized, placebo-controlled, double blinded, with four parallel groups and an equal allocation ratio in all groups. Patients 12-18 years old undergoing ﬁxed orthodontic treatment will be randomly allocated to probiotic group A (n=30) and placebo group B (n=30). Patients ≥18 years old wearing aligners (Invisalign™ ) will be randomly allocated to probiotic group C (n=30) and placebo group D (n=30). All participants will consume lozenges for one month. Assessments will be taken at baseline, at the end of the intervention and at a 2 month free-intervention follow-up. The outcome measures will be modified plaque index (PI), modified gingival index (GI) and halitosis-causing volatile sulfur compound (VSC) levels. Results will be announced at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the trial must comply with all of the following at randomization:

  * Age between 12 and 18 years for the group with conventional orthodontic appliances This age group represents the majority of patients seeking orthodontic treatment and is homogeneous regarding occupational status (high-school and lyceum students in Greece). Younger patients might present with cooperation problems.

Age ≥18 for the Invisalign™ group This age group represents the majority of patients seeking orthodontic with aligners (Invisalign™) regarding social status and other factors.

* Good general health
* Fixed orthodontic appliances Patients should have fixed labial appliances (brackets) on all teeth from central incisor to first molar, in both the maxillary and the mandibular arch. Fixed appliances should have been placed at least two months before the patient is accepted into the study and remaining treatment should be at least 3 months. All brackets will be the same (metallic, conventional/not self-ligating, same size). Molars should be banded (same bands on all molars) and all other teeth bonded.
* At least 20 natural teeth (in case of extraction orthodontic treatment patients can be enrolled two months after extractions) The outcomes will be evaluated at all teeth from first molar to first molar.

Exclusion Criteria:

* Patients will be excluded for any of the following reasons:

  * Active caries
  * Periodontitis
  * Syndromes, mental disabilities and craniofacial deformities
  * Smoking or use of other tobacco products
  * Dental fluorosis/tooth malformation
  * Antibiotics during the last 2 months
  * chlorhexidine in the previous 3 week
  * Suffering from any disease within 2 months before measurements
  * Allergy to dairy products
  * Participation in other trials Consent / assent Parents/guardians and patients will provide written informed consent and patients will provide written assent before randomization and before any procedures are applied.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Modified Silness and Löe plaque index (PI-M) | baseline-1 month
  The Silness and Löe index does not take into account the pattern of plaque accumulation in orthodontic patients. To overcome this problem, divided the tooth into mesial, distal, gingival, and incisal regions in relation to the bracket and scored plaque in each region using the four codes of the original index (0 to 3). The values are summed to obtain a total score, which ranges from 0 to 12 for each tooth. This modified index is recommended for patients with fixed orthodontic appliances because it acknowledges the usual effects of orthodontic appliances on plaque distribution and has much greater categorical discrimination.
Modified Silness and Löe plaque index (PI-M) | 1 month- 3 month
  The Silness and Löe index does not take into account the pattern of plaque accumulation in orthodontic patients. To overcome this problem, divided the tooth into mesial, distal, gingival, and incisal regions in relation to the bracket and scored plaque in each region using the four codes of the original index (0 to 3). The values are summed to obtain a total score, which ranges from 0 to 12 for each tooth. This modified index is recommended for patients with fixed orthodontic appliances because it acknowledges the usual effects of orthodontic appliances on plaque distribution and has much greater categorical discrimination.
Modified Gingival index (GI-M) | baseline-1 month
  The Gingival Index (GI) is a measure of the severity of gingivitis and is scored by measuring the amount of gingival inflammation, also considering redness and bleeding .
Modified Gingival index (GI-M) | 1 month- 3 month
  The Gingival Index (GI) is a measure of the severity of gingivitis and is scored by measuring the amount of gingival inflammation, also considering redness and bleeding.
Halitosis/ VSCs levels | baseline-1 month
  VSCs levels will recorded at each time point with the use of OralChromaTM. OralChromaTM is a portable gas chromatograph, which uses ambient air as a carrier gas and a semiconductor (In2O3) gas sensor to detect volatile sulphur compounds (VSCs), i.e. the concentrations of H2S, CH3SH and (CH3)2S.
Halitosis/ VSCs levels | 1 month- 3 month
  VSCs levels will recorded at each time point with the use of OralChromaTM. OralChromaTM is a portable gas chromatograph, which uses ambient air as a carrier gas and a semiconductor (In2O3) gas sensor to detect volatile sulphur compounds (VSCs), i.e. the concentrations of H2S, CH3SH and (CH3)2S.

CONTACTS AND LOCATIONS:
Overall Officials: Iosif Sifakakis, Associate Professor, Principal Investigator — University of Athens
Locations (1):
- National and Kapodistrian University of Athens, School of Dentistry, Departments of Orthodontics, Athens, Attica, Greece